CLINICAL TRIAL: NCT05239468
Title: A Phase 2a, Double-Blind, Randomized, Active Controlled, Parallel Group Study Evaluating the Efficacy, Safety, and Tolerability of Bezafibrate Administered in Combination With Obeticholic Acid in Subjects With Primary Biliary Cholangitis
Brief Title: Study of OCA in Combination With BZF Evaluating Efficacy, Safety and Tolerability in Participants With PBC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Intercept Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 747-214
Record Dates: First submitted 2022-01-28; First posted 2022-02-15 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Primary Biliary Cholangitis
Keywords: Primary Biliary Cholangitis; Primary Biliary Cirrhosis; Hepatic Impairment; Cirrhosis; Liver
MeSH Terms: conditions — Liver Cirrhosis, Biliary; Fibrosis | interventions — Bezafibrate; obeticholic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Double Blind (DB) Phase Treatment A: BZF 100 milligrams (mg) Immediate Release (IR) tablet (Active Comparator): Each Participant will take one OCA placebo tablet, one BZF 100 mg IR tablet and one BZF placebo tablet daily.
  Interventions: Drug: Bezafibrate 100 mg; Drug: Obeticholic Acid placebo; Drug: Bezafibrate Placebo
- Double Blind (DB) Phase Treatment B: BZF 400 mg IR tablet (Active Comparator): Each Participant will take one OCA placebo tablet and two BZF 200 mg IR tablets (to achieve 400 mg dose) daily.
  Interventions: Drug: Bezafibrate 200 mg; Drug: Obeticholic Acid placebo
- Double Blind (DB) Phase Treatment C: OCA 5 mg + BZF 100 mg IR (Experimental): Each participant will take one OCA 5 mg tablet, one BZF 100 mg IR tablet and one BZF placebo tablet, daily.
  Interventions: Drug: Bezafibrate 100 mg; Drug: Obeticholic Acid 5 mg; Drug: Bezafibrate Placebo
- Double Blind (DB) Phase Treatment D: OCA 5 mg + BZF 400 mg IR (Experimental): Each participant will take one OCA 5 mg tablet and two BZF 200 mg IR tablets (to achieve 400 mg dose) daily.
  Interventions: Drug: Bezafibrate 200 mg; Drug: Obeticholic Acid 5 mg
- Long Term Safety Extension (LTSE) Phase Treatment D of the DB phase: OCA 5 mg + BZF 400 mg IR (Experimental): Each participant will take one OCA 5 mg tablet and two BZF 200 mg IR tablets (to achieve 400 mg dose) daily.
  Interventions: Drug: Bezafibrate 200 mg; Drug: Obeticholic Acid 5 mg

INTERVENTIONS:
Drug: Bezafibrate 100 mg — One tablet of bezafibrate 100 mg IR once daily
  Arms: Double Blind (DB) Phase Treatment A: BZF 100 milligrams (mg) Immediate Release (IR) tablet; Double Blind (DB) Phase Treatment C: OCA 5 mg + BZF 100 mg IR
Drug: Bezafibrate 200 mg — Two tablets of bezafibrate 200 mg IR once daily for BZF 400 mg IR
  Arms: Double Blind (DB) Phase Treatment B: BZF 400 mg IR tablet; Double Blind (DB) Phase Treatment D: OCA 5 mg + BZF 400 mg IR; Long Term Safety Extension (LTSE) Phase Treatment D of the DB phase: OCA 5 mg + BZF 400 mg IR
Drug: Obeticholic Acid 5 mg — One tablet of obeticholic acid 5 mg tablet once daily.
  Arms: Double Blind (DB) Phase Treatment C: OCA 5 mg + BZF 100 mg IR; Double Blind (DB) Phase Treatment D: OCA 5 mg + BZF 400 mg IR; Long Term Safety Extension (LTSE) Phase Treatment D of the DB phase: OCA 5 mg + BZF 400 mg IR
Drug: Obeticholic Acid placebo — One tablet of obeticholic acid placebo tablet once daily
  Arms: Double Blind (DB) Phase Treatment A: BZF 100 milligrams (mg) Immediate Release (IR) tablet; Double Blind (DB) Phase Treatment B: BZF 400 mg IR tablet
Drug: Bezafibrate Placebo — One tablet of bezafibrate placebo tablet once daily
  Arms: Double Blind (DB) Phase Treatment A: BZF 100 milligrams (mg) Immediate Release (IR) tablet; Double Blind (DB) Phase Treatment C: OCA 5 mg + BZF 100 mg IR

SUMMARY:
Study to determine the effect of the investigational drug bezafibrate (BZF) alone and in combination with the investigational drug obeticholic acid (OCA) in participants with Primary Biliary Cholangitis (PBC).

ELIGIBILITY:
Inclusion Criteria:

* A definite or probable diagnosis of PBC
* Qualifying ALP and/or bilirubin liver biochemistry values
* Taking ursodeoxycholic acid (UDCA) for at least 12 months or no UDCA for 3 months before Day 1

Exclusion Criteria:

* History or presence of other concomitant liver diseases
* Presence of clinical complications of PBC
* History or presence of decompensating events
* Current or history of gallbladder disease
* If female, known pregnancy, or has a positive urine pregnancy test (confirmed by a positive serum pregnancy test), or lactating
* Treatment with commercially available OCA or participation in a previous study involving OCA, or other farnesoid X receptor (FXR) agonists, or peroxisome proliferator activated receptor (PPAR)-agonists within 3 months before Screening
* Unable to tolerate BZF or other fibrates, treatment with commercially available fibrates, or participation in a previous study involving fibrate within 3 months before Screening.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Change in Alkaline Phosphatase (ALP) from Baseline to Week 12 | Baseline, and at Weeks 2, 4, 6, 8, 10 and 12

SECONDARY OUTCOMES:
Change from Baseline in response rates of ≥10 percent, ≥20 percent, ≥30 percent and ≥40 percent reduction and normalization rates of biochemical disease marker ALP | Baseline and at Weeks 2, 4, 6, 8, 10 and 12
Number of participants with normalization rates of alanine aminotransferase (ALT), gamma-glutamyl transferase (GGT), alanine aminotransferase (AST), total and conjugated bilirubin and lipid panel | Baseline and at Weeks 2, 4, 6, 8, 10 and 12
Change from Baseline in biochemical disease marker GGT | Baseline and at Weeks 2, 4, 6, 8, 10 and 12
Change from Baseline in biochemical disease marker ALT | Baseline and at Weeks 2, 4, 6, 8, 10 and 12
Change from Baseline in biochemical disease marker AST | Baseline and at Weeks 2, 4, 6, 8, 10 and 12
Change from Baseline in biochemical disease markers, total & conjugated bilirubin | Baseline and at Weeks 2, 4, 6, 8, 10 and 12
Change from Baseline in lipid panel | Baseline and at Weeks 2, 4, 6, 8, 10 and 12
Change from Baseline of the plasma value of 7 alpha (α) hydroxy 4 cholesten-3 one (C4) | Baseline and at Weeks 2, 4, 6, 8, 10, and 12
Change from Baseline of the plasma value of bile acids, in unit of nanograms per milliliter (ng/ml) | Baseline and at Weeks 2, 4, 6, 8, 10, and 12

CONTACTS AND LOCATIONS:
Overall Officials: Lynda Szczech, M.D., Study Director — Intercept Pharmaceuticals, Inc
Locations (26):
- United States (17):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Southern California Gastrointestinal (GI) and Liver Centers (SCLC) - Coronado, Coronado, California
  - Facey Medical Group, Mission Hills, California
  - Schiff Center for Liver Diseases / University of Miami, Miami, Florida
  - Tampa General Medical Group, Tampa, Florida
  - Piedmont Atlanta Hospital, Atlanta, Georgia
  - Loyola University Medical Center, Maywood, Illinois
  - Ochsner Medical Center, New Orleans, Louisiana
  - Beth Israel Deaconess Medical Center Harvard Liver Research Center, Boston, Massachusetts
  - NYU Langone Medical Center, New York, New York
  - Wake Endoscopy Center, Raleigh, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Gastro One, Cordova, Tennessee
  - Gastrointestinal Associates of Northeast Tennessee, Johnson City, Tennessee
  - Methodist Clinical Research Institute (CRI), Dallas, Texas
  - Houston Methodist Cancer Center, Houston, Texas
  - American Research Corporation at the Texas Liver Institute, San Antonio, Texas
- Argentina (5):
  - Hospital Italiano La Plata, La Plata, Buenos Aires
  - DIM Clinical Privada, Ramos Mejía, Buenos Aires
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Hospital Universitario Austral, Pilar
  - Hospital Provincial del Centenario, Rosario
- Canada (3):
  - The Northern Alberta Clinical Trials and Research Centre, Edmonton, Alberta
  - Pacific Gastroenterology Associates, Vancouver, British Columbia
  - University of Montreal, Montreal, Quebec
- Azienda Ospedaliero-Universitaria di Bologna Policlinico S. Orsola-Malpighi, Bologna, Italy